CLINICAL TRIAL: NCT02699424
Title: Prospective Evaluation of 68-Ga-PSMA -PET and Early PSA Kinetics During Salvage Radiotherapy for Personalizing the Management of Men With Relapse of Prostate Cancer After Radical Prostatectomy
Brief Title: Prospective Evaluation of 68-Ga-prostate Specific Membrane Antigen (PSMA)-Positron Emission Tomograph (PET) and Early Prostatic Specific Antigen (PSA) Kinetics During Salvage Radiotherapy for Personalizing the Management of Men With Relapse of Prostate Cancer After Radical Prostatectomy
Acronym: PROPER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PP01
Record Dates: First submitted 2016-02-11; First posted 2016-03-04 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Relapsed Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Radiotherapy (Other)
  Interventions: Radiation: External radiation therapy

INTERVENTIONS:
Radiation: External radiation therapy

SUMMARY:
This is an open-label, phase II trial in patients with PSA recurrence after prostatectomy. Patients entering the study will all receive initial 50 Gray (Gy) radiotherapy (25 x 2Gy) to the prostate bed and thereafter be classified as either responders or non-responders depending on PSA response at fifth week of radiotherapy.

A 68-Ga- PSMA-PET is done before start of radiotherapy, and analyzed before fifth treatment week in order to identify cancer lesions in patients with poor PSA response. Patients with PSA response after 5 weeks of radiotherapy will not receive any subsequent therapy, whilst patients with poor PSA response may be in need for additional therapy such as radiotherapy to lymph node metastases and/or boost fractions to local recurrence. Patients with more than 3 lymph node metastases or distant metastases will not receive any more radiotherapy, but individualized systemic therapy will be started.

ELIGIBILITY:
Inclusion Criteria:

* Histological evidence of prostate cancer in the radical prostatectomy specimen
* At least 2 rising PSA values, of which the last ≥ 0.15 ng/ml
* Tumor, regional nodes, metastasis (TNM): any T, N0/x, M0/x
* Age: 18 years or older
* World Health Organization (WHO) performance status 0-1
* Life expectancy > 10 years
* Adequate laboratory findings: hematological: hemoglobin > 90 g/L (may be transfused to maintain or exceed this level) absolute neutrophil count (ANC) ≥ 1,0 x 109/L, platelets ≥ 75 x 109/L hepatic: bilirubin ≤ 1.5 x upper limit of normal (ULN), alanine aminotransferase (ALAT) ≤ 5 x ULN renal: creatinine ≤ 1.5 x ULN
* Signed written informed consent
* The patient must be able to comply with the protocol

Exclusion Criteria:

* Evidence of metastasis on imaging or in specimen (e.g. N1 at lymph-node dissection)
* Prior or ongoing treatment with hormones (antiandrogens, GnRH)
* Prior radiotherapy to the pelvis
* Previous malignancy other than prostate cancer and basalioma the past 5 years.
* Clinically significant (i.e. active) cardiovascular disease e.g. myocardial infarction (≤ 6 months), unstable angina, New York Heart Association (NYHA) grade III-IV congestive heart failure
* Severe pulmonary disease e.g. pulmonary fibrosis
* Any other serious or uncontrolled illness which in the opinion of the investigator makes it undesirable for the patient to enter the trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Tumor detection rate measured with Ga-PSMA-PET in non-responders versus responders. | PSA response is evaluated after 5 weeks of radiotherapy. Ga-PSMA-PET at baseline is compared in the PSA-responder group as compared to the non-responder group
Assessment of PSA response during radiotherapy. | Is evaluated once weekly during radiotherapy, duration of radiotherapy is 35 days; 70 Gy in 2 Gy fractions.

OTHER OUTCOMES:
Assessment of PSA response post treatment. | Is evaluated at 6, 12, 24, and 60 months post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Adalsteinn Gunnlaugsson, MD, PhD, Principal Investigator — Lund University Hospital, Department of Oncology
Locations (1):
- Lund University Hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gunnlaugsson A, Johannesson V, Wieslander E, Brun E, Bitzen U, Stahl O, Bratt O, Ahlgren G, Ohlsson T, Kjellen E, Nilsson P. A prospective phase II study of prostate-specific antigen-guided salvage radiotherapy and 68Ga-PSMA-PET for biochemical relapse after radical prostatectomy - The PROPER 1 trial. Clin Transl Radiat Oncol. 2022 Jul 5;36:77-82. doi: 10.1016/j.ctro.2022.07.001. eCollection 2022 Sep. PMID 35873652